CLINICAL TRIAL: NCT06580990
Title: Effectiveness of a Telerehabilitation Programme Based on Specific Neck Specific Neck Exercises in Patients With Whiplash-associated Disorders. Randomised Clinical Trial Controlled and Multicentric
Brief Title: Neck-specific Exercises Effectively Improves Whiplash-associated Disorders.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Concepcion (Other)
Responsible Party: Principal Investigator, Mario Muñoz Bustos, Associate professor, Universidad de Concepcion
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBB 1682-2024
Record Dates: First submitted 2024-08-26; First posted 2024-08-30 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Whiplash-associated Disorders
Keywords: Whiplash; Exercise; Pain; Disability; Telerehabilitation
MeSH Terms: conditions — Whiplash Injuries; Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: This study will be a single-blinded, randomised, controlled clinical trial and multicentric
Who Masked: Outcomes Assessor
Masking Description: the evaluator does not have access to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Specific neck exercises with the Spinetrack (Experimental): Exercise the deep neck muscles using the Spinetrak twice a week for 6 weeks.
  Interventions: Procedure: specific neck exercises with the Spinetrack
- Standard specific neck exercises (Active Comparator): Exercise programme for the deep neck musculature twice a week for 6 weeks.
  Interventions: Procedure: specific neck exercises
- Usual care group (No Intervention): This group will receive instructions from the doctor based on their assessment, taking into account education and analgesics

INTERVENTIONS:
Procedure: specific neck exercises with the Spinetrack — This group will receive an telerehabilitation exercise programme for the deep neck musculature using the spinetrack
  Other Names: SES
  Arms: Specific neck exercises with the Spinetrack
Procedure: specific neck exercises — This group will receive a telerehabilitation programme with exercise for the deep neck musculature
  Other Names: SSE
  Arms: Standard specific neck exercises

SUMMARY:
Whiplash-associated disorders (WAD) are common injuries from motor vehicle accidents, typically treated with a return to normal activity and neck exercises. The Spinetrack device has been approved for deep neck musculature training, but its impact on pain and disability in subacute WAD patients in a virtual setting hasn't been evaluated yet. This study aims to assess the effect of a telerehabilitation programme using the Spinetrack device on pain and self-perceived disability in subacute WAD I and II patients. The single-blinded, randomised, controlled clinical trial will involve 102 participants divided into three groups: a telerehabilitation group using Spinetrack, a group with a standard telerehabilitation programme, and a usual care group. Training will be conducted via video call for six weeks. The study expects to confirm that deep neck musculature training reduces pain and disability in WAD patients and establish Spinetrack as an efficient tool for subacute WAD treatment.

DETAILED DESCRIPTION:
Introduction: Whiplash-associated disorders (WAD) are a group of clinical manifestations experienced by individuals following a sudden acceleration-deceleration mechanism of the neck. WAD are the most common injuries resulting from a motor vehicle accident. The mainstays of WAD treatment are a return to normal activity and both general and deep neck musculature exercises. Recently, a device called Spinetrack has been validated to facilitate training of the deep craniocervical musculature. This device can even be adapted for use in a virtual format. However, to date, it has not been determined how this device contributes to the improvement of pain and disability in individuals with subacute WAD in a virtual context.

Objective: The aim of this study is to evaluate the effect of a telerehabilitation programme, which is based on specific neck exercises with the Spinetrack, on pain and self-perceived disability in people with WAD I and II in the subacute stage.

Methods: This study is a single-blinded, randomised, controlled clinical trial. A total of 102 subjects with WAD I and II will be recruited according to the Quebec Task Force classification in the subacute stage. The participants will be randomised into three groups: a telerehabilitation group based on specific neck exercises with the Spinetrack (SES), a treatment group with a telerehabilitation programme with standard specific neck exercises (SSE), and a usual care group (UCG).

Training will be carried out via video call over 12 sessions distributed over six weeks, with two sessions per week. The main outcome variables will be pain and perceived disability.

Expected Results: The investigators anticipate that training the deep neck musculature will reduce pain and disability in patients with WAD. It is expected to demonstrate the device's function as a tool for self-management of neck symptoms and to provide the health care system with an efficient device for the treatment of subacute WAD.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-65 years
* Patients with WAD, defined as cervical pain or disability resulting from a resulting from a collision or similar trauma, grade I-II according to QTF8 in subacute stage from 7 days to 12 weeks.
* Have internet connection and a device to communicate (telephone, television, computer).
* NPRS up to moderate category (4 out of 10).38
* IDC score up to moderate category (15 out of 50).

Exclusion Criteria:

* Screening for cervical fractures ruled out by the National Emergency X-ray Utilization Study (NEXUS) criteria. (Focal neurological deficits such as paralysis, paraesthesia, speech, vision or hearing impairment; Midline spinal cord tenderness; Altered spinal cord level Altered level of consciousness; Intoxication; Distraction injury defined as a serious injury to another part of the body; or other serious injury to another part of the body that could distract from the neck injury).
* Previous cervical spine, jaw and upper extremity surgeries
* Traumatic brain injury
* Neck pain and disability from abuse, domestic violence or fights
* Difficulty hearing and understanding instructions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Pain intensity as measured by Numeric Pain Rating Scale (NPRS) | Baseline, at 6 and 12 weeks
  NPRS is a validated instrument assessing average pain intensity over the past 24 hour period. Possible scores range from 0 (no pain) to (wort possible pain).
Disability as measured by Neck disability Index (NDI) | Baseline, at 6 and 12 weeks
  This questionnaire has been validated to give information as to how the neck pain has affected the ability to manage in everyday life.The original report provided scoring intervals for interpretation, as follows: 0 to 4 = no disability 5 to 14 = mild 15 to 24 = moderate 25 to 34 = severe Above 34 = complete.

SECONDARY OUTCOMES:
Global Perceived Effect as measured by Global Perceived Effect Scale (-7 to +7 Likert Scale) | Baseline, at 6 and 12 weeks
  The GRoC is a single-item, recall-based questionnaire of well-being that is based on progress (or lack of progress) since an initial treatment encounter. Patients are routinely asked to make global ratings on changes in regards to their level of well-being since the previous week's treatment on a 15-point self-report scale (from -7 to 7)
Self-perception of vestibular difficulty as measured by Dizziness Handicap Inventory (DHI) | Baseline, at 6 and 12 weeks
  The DHI is a 25-item self-reported measure with three categories: functional, emotional, and physical. The patient rates their perceived disability due to their dizziness by answering each question with - yes, sometimes, or no.
dizziness induced by dynamic visual input as measured by Visual vertigo analogue scale (VVAS) | Baseline, at 6 and 12 weeks
  Vertigo symptoms that are triggered by visual stimuli. Scale have 9 items and each one is answered from 0 (no vertigo) to 10 (maximum vertigo).
Impact of headaches on daily life Headache intensity as measured by The Headache Impact Test (HIT-6) | Baseline, at 6 and 12 weeks
  HIT-6 is a questionnaire for measuring the impact of headache. A total of six questions are completed by the patient. They focus on daily activities such as work, education, home situation and leisure time. The HIT-6 gives a general overview of the impact of headache, including pain intensity, impairment and other items. A higher score corresponds to higher impact.
Fear or excessive aversion to physical movement or exercise, also called kinesiophobia as measured by Tampa Scale of Kinesiophobia (TSK) | Baseline, at 6 and 12 weeks
  The TSK is a 17 item assessment checklist. It uses a 4-point Likert scale (Strongly Disagree-Disagree-Agree-Strongly Agree) with statements that have been later linked to the model of fear-avoidance, fear of work-related activities, fear of movement, and fear of re-injury
depression and anxiety as measured by Hospital Anxiety and Depression Scale (HADS) | Baseline, at 6 and 12 weeks
  The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21)
Difficulties people sometimes have after stressful life events as measured by Impacto of event scale (IES) | Baseline, at 6 and 12 weeks
  Post-traumatic stress disorder (PTSD) symptoms. Event Impact Scale-Revised has 22 items and 3 subscales: Intrusion, Avoidance and Hyperarousal. It uses a Likert-type scale to evaluate the intensity of the of the symptomatology (0,1,2,2,3,4. From 'Not at all' to 'Extremely').
  to 'Extremely')
Measures the somatic and emotional symptoms common to central sensitization syndrome (CSS) as measured by the Central Sensitization Inventory (CSI) | Baseline, at 6 and 12 weeks
  Pathophysiologic process in which the central nervous system undergoes changes that alter its processing of pain and other sensory stimuli, may be the mechanism underlying various conditions in which patients have unexplained pain and fatigue. The CSI consists of two parts; Part A includes 25 questions related to common CSS symptoms. Part B determines if the patient has been diagnosed with certain CSS disorders or related disorders, such as anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Muñoz Bustos, MSc, Principal Investigator — Universidad de Concepcion
Locations (1):
- Universidad de Concepción, Concepción, Región del Biobío, Chile

IPD SHARING:
Plan to Share IPD: No